CLINICAL TRIAL: NCT06015685
Title: Embedding and Evaluating Multidisciplinary Diabetes Management and Continuous Glucose Monitoring Into Primary Care for a Vulnerable Population
Brief Title: Embedded Primary Care MultiDisciplinary Diabetes Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Center for Diabetes Translation Research (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Diabetes Association (Other)
Responsible Party: Principal Investigator, Britt A. Marshall, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006033; P30DK111024 (NIH)
Record Dates: First submitted 2023-08-22; First posted 2023-08-29 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Primary Care; Continuous Glucose Monitoring (CGM); Diabetes Management; Multidisciplinary care
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Embedded clinic at Midtown (Experimental): Using the Emory Clinical Data Warehouse (CDW), all patients of Emory Primary Care Midtown with HbA1c >9% who are not currently under the care of an endocrinologist or the diabetes management program at Emory will be invited to participate in this embedded DM management clinic.
  Interventions: Other: Embedded Clinic
- Routine Care- Dunwoody Family Medicine Clinic (Other): The control population will be drawn using electronic health record data of diabetes patients at Dunwoody Family Medicine Clinic. Information from the Electronic Health Record will be de-identified after extraction. Control participants will be frequency matched.
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Embedded Clinic — Once a week, a Primary Care clinic half-day will be dedicated to multi-disciplinary, team-based DM care. The inter-professional team will include an Internal Medicine attending physician, an Internal Medicine resident, a DM educator, a nurse trained in professional CGM, a behavioral health provider, and a social worker to assist in finding resources for housing, food, and patient assistance programs.
  Other Names: multi-disciplinary, team-based DM care
  Arms: Embedded clinic at Midtown
Other: Routine Care — Researchers will use a 2:1 ratio of control to intervention patients. Using the CDW, researchers will identify a control population [patients who receive routine care (i.e., referral to subspecialty care)], who will be a propensity-matched cohort of individuals with similar age, gender, race/ethnicity, zip codes, insurance type, visit dates, and co-morbidities (Charlson Comorbidity Index) as the intervention group.
  Other Names: Control Group
  Arms: Routine Care- Dunwoody Family Medicine Clinic

SUMMARY:
The purpose of this study is to improve diabetes management for patients at Midtown General Internal Medicine Clinic (Aim 1). The clinic offers dedicated diabetes care on certain days with trained providers able to offer dedicated diabetes care. The clinic will also make sure to address other aspects of life and health that may impact an individual's ability to manage their diabetes - food insecurity, housing insecurity, knowing about healthy food, finding ways to exercise, and mental health. The study will also train the medical residents to be able to participate in this dedicated diabetes care (Aim 2).

DETAILED DESCRIPTION:
There is a widening quality of care gap in diabetes mellitus (DM) management that sees Black and Hispanic patients with much higher rates of DM complications and hospitalizations compared to their white counterparts. Primary Care is the frontline for DM prevention and management; however, Primary Care Clinics, including Internal Medicine resident continuity clinics, struggle to improve DM metrics. The lack of resources, such as time and personnel, is a significant limiting factor in strategies that would allow these clinics to optimize care. As a result, the current DM management model was created, in which Primary Care providers refer patients with elevated hemoglobin A1c (HbA1c) to subspecialty care. This process is inefficient, overwhelms subspecialty practices, and most importantly does not address the social determinants of health that often make it difficult for patients to get their DM under control.

This traditional model also comes with a potential institutional financial cost. There is a perception that reducing upfront costs of care can make a system more economically viable; yet this can have devastating results for a system and for its patients on the back end. For example, HbA1c is a Merit-based Incentive Payment System Clinical Quality Measure if a patient population is not supported in their efforts for DM control, this can translate to monetary loss annually for the Emory Healthcare System. In addition, there are also potential losses to the system related to long-term morbidity and mortality risks of elevated HbA1c over time.

Studies have shown that a multi-disciplinary approach including physician, dietitian, DM education, psychotherapy, and social work services functioning concurrently and cooperatively has the potential to positively change the current paradigm. Given the vital role Primary Care plays in the management of all aspects of patient care, including physical and psychosocial well-being, this care delivery model is optimally designed to have the most impact and success in the Primary Care Clinic setting. The research team proposes to embed a multi-disciplinary diabetes-focused clinic within Primary Care in the Emory Healthcare System where this approach would create a central location for all the patients' DM needs, provide efficient care that helps patients address social and economic barriers, and engage the care team through between-clinic touchpoints to motivate patients to take agency over their health. This also provides a venue to implement modern technologies for DM management, such as continuous glucose monitoring (CGM). Despite its proven efficacy in DM management, CGM remains an understudied intervention in Primary Care, especially in patient populations that would otherwise have difficulty accessing specialty care. Researchers anticipate that these changes will enable improved adherence to follow-up visits and treatment.

In addition to the benefits of streamlined patient care, this model also offers the opportunity to enhance Internal Medicine residency education. Investigators intend to develop a hybrid clinical/educational curriculum for residents that capitalizes on and models appropriate resource utilization through an integrated care model and provides early exposure to multi-disciplinary care and CGM.

ELIGIBILITY:
Aim 1 (Embedded diabetes clinic):

Inclusion Criteria:

* Age 18+
* Patient at Midtown Diabetes Clinic
* Able to consent
* HbA1c >=9%

Exclusion Criteria:

* Not planning to follow up at Midtown
* Pregnancy
* Followed by Endocrinology as a specialist

Aim 2 (Embedded diabetes clinic and curriculum):

Inclusion Criteria:

- All residents in Midtown Primary Care are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of embedded clinic patients with an HbA1c >9% | Baseline and 6 months
  Percentage of participants with HbA1c >9% since the embedded clinic implementation. Data will be assessed from electronic medical records (EMR)
Change in acceptability of intervention measure (AIM) | Baseline and 6 months
  AIM score is a four-item measures of implementation outcomes that are often considered "leading indicators" of implementation success (likert scale 1-5 with 5 being best outcome) at the baseline and 6-month follow-up visits will be used by the team members to assess the acceptability of model implementation.
Change in feasibility of intervention measure (FIM) scores | Baseline and 6 months
  FIM score is a four-item measures of implementation outcomes that are often considered "leading indicators" of implementation success likert scale 1-5 with 5 being best outcome) at the baseline and 6-month follow-up visits will be used by the team members to assess the feasibility of model implementation.

SECONDARY OUTCOMES:
Change in weight | Baseline, 3 months, and 6 months
  Change in weight will be assessed from available measurements in EMR.
Change in body mass index (BMI) | Baseline, 3 months, and 6 months
  BMI will be calculated from available measurements in EMR
Change in diabetes self-efficacy score | Baseline, 3 months, and 6 months
  Participants will complete the diabetes management self-efficacy scale (DMSES). It assesses the extent to which respondents are confident they can manage their blood sugar, diet, and level of exercise. Responses are rated on a 5-point scale ranging from ''can't do at all'' to ''certain can do'' (1, 5). In this scale, higher scores indicate higher self-efficacy in performing Diabetes self-management (DSM) activities.
Change in depression status | Baseline, 3 months, and 6 months
  The 9-question Patient Health Questionnaire (PHQ9) is a diagnostic tool to screen adult patients in a primary care setting for the presence and severity of depression. Scores represent: 0-5 = mild 6-10 = moderate 11-15 = moderately severe. 16-20 = severe depression.
Change in the patient-reported quality of life score | Baseline, 3 months, and 6 months
  Participants will complete the Patient-Reported Outcomes Measurement Information System (PROMIS) survey. The possible score ranges from 0 to 20 points in each case. 0 points represent the patient's most severe physical and/or mental impairment, while 20 points represent the best possible state of health.
Change in anxiety score | Baseline, 3 months, and 6 months
  Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. Scores represent 0-4: Minimal Anxiety; 5-9: Mild Anxiety; 10-14: Moderate Anxiety; a score greater than 15: Severe Anxiety
Change in food insecurity | Baseline, 3 months, and 6 months
  Participants will complete the Latin American and Caribbean (ELSCA) Household Food Security Measurement Scale. This scale uses a set of 15 questions, with yes/no response categories, seven of which are for households with children. Each question asks the respondent whether he/she or any other household member has experienced a certain manifestation of food insecurity in the previous three months. Households that affirm 3 items are classified as food insecure.
Change in Housing Insecurity | Baseline, 3 months, and 6 months
  Percentage of participants of being at risk for housing insecurity by answering the 2-question housing insecurity instrument: (1) "Are you worried or concerned that in the next 2 months you may not have stable housing that you own, rent, or stay in as part of a household?" with responses of "yes" or "no," and (2) "How likely do you think it would be that you would have to use a homeless shelter in the next 6 months?" with 4 response options ranging from "very unlikely" to "very likely."
Change in urine microalbumin | Baseline, 3 months, and 6 months
  Change in urine microalbumin (mcg/mg min 0 and higher the worse the outcome) will be calculated from available laboratory assessments from EMR

CONTACTS AND LOCATIONS:
Overall Officials: Britt A Marshall, MD, Principal Investigator — Emory University
Locations (1):
- Emory Primary Clinic Care at Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share deidentified individual participant's data that underlie the results reported in the article after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The research team will share the deidentified data immediately following publication, with no known end date.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims specified in their proposal
  All proposals should be sent to britt.marshall@emory.edu.

DOCUMENTS (1):
  • Informed Consent Form (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT06015685/ICF_000.pdf